CLINICAL TRIAL: NCT02433301
Title: PET/MR-imaging and Circulating Tumour Cells to Evaluate the Response of Chemotherapy in Patients With Gastroesophageal Junction Cancer
Brief Title: PET/MR-imaging to Differentiate Between Responders and Non-responders Receiving Preoperative Chemotherapy
Status: Completed | Type: Observational
Sponsor: Rikshospitalet University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Belmouhand, Medical student, Rikshospitalet University Hospital
Other Study IDs: H-1-2014-076
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Gastroesophageal Junction Cancer
Keywords: chemotherapy; GEJ cancer; PET/MR-imaging

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — Four biopsies from each patient harvested from the Gastroesophageal junction cancer

SUMMARY:
The incidence of malignity in the gastroesophageal junction (GEJ) is rising in Denmark, 400 new cases annually 1. 60% of the patients with GEJ cancer have disseminated disease (M1-stage) at time of diagnosis and are consequently unable to undergo curative intended surgery. The prognosis is poor, with 5-year survival rates of approximately 2 % for these 60% and the treatment only consists of palliative therapy 1. For the remaining approximately 40 % who are assessed as candidates for curative intended surgery, the 5-year survival rate is 33 % 1. This emphasizes the need for further research and knowledge concerning tumour biology and spontaneous course of the disease.

In Denmark, all cancer patients are enrolled in a specific cancer program. The primary diagnostic work-up for GEJ cancers includes gastroscopy with biopsy, blood samples, ultrasonography scan, Positronemissionstomography (PET) and Computed tomography (CT) alone or PET/CT in combination 2. From these parameters physicians determine resectability and TNM-stage (tumour staging), which is substantial for the prognosis and future treatment. The primary goal is to achieve a macroscopically resection of tumour and lymphnodes in relation to the stomach and oesophagus (Esophagectomi a.m. Ivor Lewis and D1+ lymphadenectomy in the abdomen and thorax). In addition to surgery, patients receive perioperative chemotherapy, which consist of three series of chemotherapy preoperative and three series postoperative approximately 21-28 days after surgery.

Approximately 12.6 % of patients receiving perioperative chemotherapy prior to surgery will have disease progression due to chemotherapy resistance during the therapy 3. This unintentionally leads to shifting these patients from the resectable group to non-resectable group (palliative treatment). Thus, the possibility for detecting response to perioperative chemotherapy is of great interest. A paradigm shift towards an individualised tailored therapy form has emerged in recent years, which potentially require a higher need for diagnosis on molecular level. Today most molecular biological methods apply tissue samples for in-vitro analyses, but new radiological tools provide opportunity for non-invasive examinations; for example PET can with a radioactive sugar compound: Flour-18 deoxyglucose (18F-FDG). This compound is injected through a catheter in a larger vein (media cubiti vein) and absorbed in cells with increased metabolism - especially cancer cells. A PET scanner registers the absorption; this radiology modality can provide valid information, which is essential for non-invasive tumour staging and monitoring response under a specific therapy.

A new diagnostic modality is PET scan combinated with magnetic resonance (PET/MR) simultaneously. So far, no studies have conducted an evaluation of simultaneous PET/MR scan to assess the perioperative chemotherapy response in patients with GEJ cancer. However, some studies suggest that commercially available PET/MR scanner might contribute in a diagnostic elucidation 6. Simultaneous PET/MR scan might in theory minimize the misinterpretations of potential response changes after chemotherapy, which can appear in the interval between separate PET, CT and MR scans 4,5,7. Studies have found PET scan of GEJ cancer could be helpful as a prognostic tool to differentiate between responders and non-responders during chemotherapy 9. Standardized uptake value (SUV) is a unit that display the absorption of 18F-FDG and is used routinely to quantify tumour glucose metabolism in PET scan 8. A change of more than 35 % in SUV measurements before and after the induction of chemotherapy is considered as the definition of responders and non-responders in earlier studies 9.

The MR technique is based on magnetic fields and radio waves. Diffusion Weighted Imaging (DWI) is a non-invasive MR-modality, which measures the changes in water diffusion (Brownian movements) throughout tissue. These changes are measured in Apparent Diffusion Coefficient (ADC), a parameter derived from DWI and reflects the change in diffusion 7. ADC and DWI can be used to differentiate between benign and malignant tumours, due to a larger cell density in malignant tumours. Consequently, malignant tissue has a decreased diffusion relative to normal tissue. ADC has been used as a factor in some studies to predict the response to chemotherapy 10. A single study has shown a rise in ADC-value two weeks after initiation of chemotherapy in patients with GEJ cancer, and demonstrated that the percentage change in ADC-value between the groups (responders and non-responders) is significantly different 11. Simultaneous PET- and MR scan might be very useful to evaluate the response to chemotherapy in patients with GEJ cancer compared with these parameters alone. The opportunity for a more individualised tailored treatment in future might be possible with PET/MR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically verified adenocarcinoma of the Gastroesophageal junction and assessed as operable.

Exclusion Criteria:

* Under 18 of age
* Not given informed consent
* Other histological cancers besides adenocarcinoma
* Metal in the body that would contraindicate MR-imaging
* Allergies for contrast
* Claustrophobia
* Not a candidate for perioperative chemotherapy and surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to the Department of Surgical Gastroenterology, Rigshospitalet, with histologically verified adenocarcinoma of the Gastroesophageal junction and assessed as operable. Informed consent is required from each patient
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To Study wether molecular PET/MR-imaging can measure a significant difference between responders and non-responders receiving perioperative chemotherapy | 8 Months

SECONDARY OUTCOMES:
To examine if DWI and ADC can identify lymph nodes suspected for malignancy and correlate these with findings from the resected tumour preparation | 8 Months
To correlate a possible difference in responders and non-responders to survival, disease progression prior to surgery, inoperability, surgical complications and tolerance of both preoperative- and postoperative chemotherapy | 8 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Larsen AC, Hollander C, Duval L, Schonnemann K, Achiam M, Pfeiffer P, Yilmaz MK, Thorlacius-Ussing O, Baeksgaard L, Ladekarl M. A nationwide retrospective study of perioperative chemotherapy for gastroesophageal adenocarcinoma: tolerability, outcome, and prognostic factors. Ann Surg Oncol. 2015 May;22(5):1540-7. doi: 10.1245/s10434-014-4127-2. Epub 2014 Oct 28. PMID 25348777
- [Background] Gambhir SS. Molecular imaging of cancer with positron emission tomography. Nat Rev Cancer. 2002 Sep;2(9):683-93. doi: 10.1038/nrc882. PMID 12209157
- [Background] Basu S, Alavi A. Unparalleled contribution of 18F-FDG PET to medicine over 3 decades. J Nucl Med. 2008 Oct;49(10):17N-21N, 37N. No abstract available. PMID 18832112
- [Background] Thoeny HC, Ross BD. Predicting and monitoring cancer treatment response with diffusion-weighted MRI. J Magn Reson Imaging. 2010 Jul;32(1):2-16. doi: 10.1002/jmri.22167. PMID 20575076
- [Background] Jadvar H, Colletti PM. Competitive advantage of PET/MRI. Eur J Radiol. 2014 Jan;83(1):84-94. doi: 10.1016/j.ejrad.2013.05.028. Epub 2013 Jun 18. PMID 23791129
- [Background] Rakheja R, Chandarana H, DeMello L, Jackson K, Geppert C, Faul D, Glielmi C, Friedman KP. Correlation between standardized uptake value and apparent diffusion coefficient of neoplastic lesions evaluated with whole-body simultaneous hybrid PET/MRI. AJR Am J Roentgenol. 2013 Nov;201(5):1115-9. doi: 10.2214/AJR.13.11304. PMID 24147485
- [Background] Zhu W, Xing L, Yue J, Sun X, Sun X, Zhao H, Yu J. Prognostic significance of SUV on PET/CT in patients with localised oesophagogastric junction cancer receiving neoadjuvant chemotherapy/chemoradiation:a systematic review and meta-analysis. Br J Radiol. 2012 Sep;85(1017):e694-701. doi: 10.1259/bjr/29946900. Epub 2012 Feb 14. PMID 22337686
- [Background] Padhani AR, Liu G, Koh DM, Chenevert TL, Thoeny HC, Takahara T, Dzik-Jurasz A, Ross BD, Van Cauteren M, Collins D, Hammoud DA, Rustin GJ, Taouli B, Choyke PL. Diffusion-weighted magnetic resonance imaging as a cancer biomarker: consensus and recommendations. Neoplasia. 2009 Feb;11(2):102-25. doi: 10.1593/neo.81328. PMID 19186405
- [Background] Weber MA, Bender K, von Gall CC, Stange A, Grunberg K, Ott K, Haberkorn U, Kauczor HU, Zechmann C. Assessment of diffusion-weighted MRI and 18F-fluoro-deoxyglucose PET/CT in monitoring early response to neoadjuvant chemotherapy in adenocarcinoma of the esophagogastric junction. J Gastrointestin Liver Dis. 2013 Mar;22(1):45-52. PMID 23539390